CLINICAL TRIAL: NCT03722823
Title: An Open-label, Non-randomized, Single-dose, Parallel-group, Safety, Tolerability, and Pharmacokinetic Study of Tucatinib Administered at 300 mg in Fasted, Hepatically-impaired Male and Female Subjects and Fasted Matched-control Healthy Subjects
Brief Title: A Safety Study of Tucatinib in Healthy and Hepatically-Impaired Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONT-380-009
Record Dates: First submitted 2018-10-24; First posted 2018-10-29 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — tucatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: Healthy (Active Comparator): Match-controlled healthy subjects with normal hepatic function
  Interventions: Drug: Tucatinib
- Group 2: Mild Hepatic Impairment (Experimental): Subjects with Mild hepatic impairment (Child-Pugh Class A, score of 5 or 6)
  Interventions: Drug: Tucatinib
- Group 3: Moderate Hepatic Impairment (Experimental): Subjects with Moderate hepatic impairment (Child-Pugh Class B, score of 7 to 9)
  Interventions: Drug: Tucatinib
- Group 4: Severe Hepatic Impairment (Experimental): Subjects with Severe hepatic impairment (Child-Pugh Class C, score of 10 to 14)
  Interventions: Drug: Tucatinib

INTERVENTIONS:
Drug: Tucatinib — 300mg oral single dose

SUMMARY:
The investigators are doing this study to find out if tucatinib is safe for patients with liver problems. This study will look at participants with mild, moderate, and severe liver problems. For each participant with liver problems who takes part, a matching healthy participant who is of similar age, similar body mass index (BMI), and of the same sex will also take part. The study will look at how the drug affects healthy participants compared to participants with liver problems.

DETAILED DESCRIPTION:
This study is being conducted to provide information to develop dosing recommendations for tucatinib in subjects with hepatic impairment. The current study will be carried out in subjects with hepatic impairment according to 3 different Child-Pugh (CP) categories (Mild, Moderate, and Severe impairment), and in matched-control healthy subjects. The minimum number of matched-control healthy subjects will be enrolled in order to ensure that each hepatically-impaired subject has a healthy match. Each matched-control healthy subject will be enrolled following the enrollment of a Mild and/or Moderate and/or Severe hepatic impairment subject and will be matched by age (+/- 10 years), by BMI (+/- 20%), and by sex to the enrolled hepatic impairment subject(s). Each healthy subject may be matched with up to 1 subject within each hepatic impairment group. Based on these criteria, with 3 cohorts of 8 hepatically-impaired subjects enrolled in the study, the number of healthy control subjects required to be enrolled will be at least 8 and not more than 24.

ELIGIBILITY:
Inclusion Criteria:

* In good general health, except for additional inclusion criteria related to subjects with hepatic impairment
* Within body mass index (BMI) range of 18 to 37 kg/m^2 (inclusive)
* Males capable of fathering a child must agree to use contraception from check in through 90 days after dose administration
* Females must be of nonchildbearing potential
* Able to understand and provide written informed consent
* Able to comply with all study procedures, including the 3-night stay at the clinical site and follow-up phone call
* Healthy subjects only: matched to subjects with Mild and/or Moderate and/or Severe hepatic impairment in sex, age (+/- 10 years), and BMI (+/- 20%).
* Hepatic impairment subjects only: considered to have Mild, Moderate, or Severe hepatic impairment that has been clinically stable for at least 1 month
* Hepatic impairment patients only: currently on stable medication regimen

Exclusion Criteria:

* Subjects with at-rest vital signs outside of the following ranges: heart rate (40 to 120 bpm), systolic blood pressure (90 to 150 mmHg), diastolic blood pressure (40 to 95 mmHg)
* Clinically significant abnormal laboratory values or physical examination findings
* Evidence/history of long QT syndrome
* Use of drugs/substances known to be inhibitors or inducers of CYP3A4 or CYP2C8 enzyme within 30 days
* Consumption of foods or beverages containing poppy seeds, grapefruit, or Seville oranges within 7 days of check-in
* Consumption of alcohol-, citric acid-, caffeine-, or xanthine-containing foods or beverages within 48 hours prior to check in
* Subjects with known alcohol and/or drug abuse within 1 month prior to check in
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance
* History of congenital nonhemolytic hyperbilirubinemia
* History of stomach or intestinal surgery that would potentially alter absorption and/or excretion of orally administered drugs
* Prior doses of tucatinib
* Prior dose of any investigational drug within the past 30 days or 5 half-lives

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | Up to 48 hours
  Pharmacokinetic (PK) endpoint of tucatinib
Time of maximum observed concentration (Tmax) | Up to 48 hours
  PK endpoint of tucatinib
Area under the concentration-time curve (AUC) from time 0 to the last quantifiable concentration (AUC[0-t]) | Up to 48 hours
  PK endpoint of tucatinib
AUC from time 0 to infinity (AUC[0-inf]) | Up to 48 hours
  PK endpoint of tucatinib
Percentage extrapolation for AUC (%AUCextrap) | 48 hours
  PK endpoint of tucatinib
Apparent terminal elimination rate constant (λz) | Up to 48 hours
  PK endpoint of tucatinib
Apparent terminal elimination half-life (t½) | Up to 48 hours
  PK endpoint of tucatinib
Apparent total clearance | Up to 48 hours
  PK endpoint of tucatinib
Apparent volume of distribution during the terminal phase | Up to 48 hours
  PK endpoint of tucatinib
Mean residence time (MRT) | Up to 48 hours
  PK endpoint of tucatinib

SECONDARY OUTCOMES:
Cmax | Up to 48 hours
  PK endpoint of ONT-993
Tmax | Up to 48 hours
  PK endpoint of ONT-993
AUC[0-t] | Up to 48 hours
  PK endpoint of ONT-993
(AUC[0-inf]) | Up to 48 hours
  PK endpoint of ONT-993
%AUCextrap | Up to 48 hours
  PK endpoint of ONT-993
λz | Up to 48 hours
  PK endpoint of ONT-993
t½ | Up to 48 hours
  PK endpoint of ONT-993
MRT | Up to 48 hours
  PK endpoint of ONT-993
Incidence of adverse events (AEs) | Up to 9 days
  As determined by assessment of AEs, clinical laboratory tests, physical examinations, vital signs measurements, and 12-lead ECG

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Woolery, PharmD, BCOP, Study Director — Seagen Inc.
Locations (4):
- United States (4):
  - Orange County Research Center, Tustin, California
  - Orlando Clinical Research Center, Orlando, Florida
  - NOCCR Knoxville and Volunteer Research Group, Knoxville, Tennessee
  - Texas Liver Institute, San Antonio, Texas

REFERENCES:
- [Derived] Topletz-Erickson AR, Lee AJ, Mayor JG, Sun H, Abdulrasool LI, Rustia EL, Walker LN, Endres CJ. The Pharmacokinetics and Safety of Tucatinib in Volunteers with Hepatic Impairment. Clin Pharmacokinet. 2022 Dec;61(12):1761-1770. doi: 10.1007/s40262-022-01183-6. Epub 2022 Dec 5. PMID 36471222